CLINICAL TRIAL: NCT03610386
Title: In Vitro Study Of the Effects of the Menthoxypropanediol, an Anti-TRPM8, in the Atopic Dermatitis Pruritus
Brief Title: Effects of an Anti-TRPM8 in the Atopic Dermatitis Pruritus
Acronym: DA-TRPM8
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Collaborators: Beiersdorf (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DA-TRPM8 (29BRC18.0077)
Record Dates: First submitted 2018-06-12; First posted 2018-08-01 (Actual); Last update posted 2021-12-28 (Actual); Status verified 2021-12

CONDITIONS: Atopic Dermatitis
Keywords: Atopic; Dermatitis; TRPM8; menthol
MeSH Terms: conditions — Dermatitis, Atopic; Dermatitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Two biopsies of skin (4 mm diameter each) will be taken under local anesthetic in the service of dermatology of Brest CHRU. They will be situated in a pruritic lesion area little or not visible (inside of the arm, the back …).One of two biopsies will be left in culture for 24 hours and then the biopsy will be cut in half: half will be used for immunohistochemical analyzes, the second half for transcriptomic analyzes .
  Interventions: Other: No adding menthoxypropanediol to the biopsy
- Treatment with menthoxypropanediol (Experimental): Two biopsies of skin (4 mm diameter each) will be taken under local anesthetic in the service of dermatology of Brest CHRU. Thy will be situated in a pruritic lesion area little or not visible (inside of the arm, the back …).One of two biopsies will be left in culture for 24 hours. Then the menthoxypropanediol (200 µM) will be applied topically on this explant and left for 6 hours. Then the biopsy will be cut in half: half will be used for immunohistochemical analyzes, the second half for transcriptomic analyzes.
  Interventions: Other: Adding menthoxypropanediol to the biopsy

INTERVENTIONS:
Other: Adding menthoxypropanediol to the biopsy — Two biopsies of skin (4 mm diameter each) will be taken under local anesthetic in the service of dermatology of Brest CHRU. They will be situated in a pruritic lesion area little or not visible (inside of the arm, the back …). One of the two biopsies will receive menthoxypropanediol topically.
  Arms: Treatment with menthoxypropanediol
Other: No adding menthoxypropanediol to the biopsy — Two biopsies of skin (4 mm diameter each) will be taken under local anesthetic in the service of dermatology of Brest CHRU. They will be situated in a pruritic lesion area little or not visible (inside of the arm, the back …). One of the two biopsies will not receive menthoxypropanediol.
  Arms: Control

SUMMARY:
The aim of the study is to analyse the effect of the menthoxypropanediol, a derivative of menthol, on the pruritus of atopic dermatitis (ex vivo study).

DETAILED DESCRIPTION:
AD is a fairly common pathology whose prevalence in Western Europe and the United States is estimated at 10 to 15% in children and 4 to 7% in adults. This frequency has been steadily increasing for several decades. However, while the prevalence is increasing rapidly in emerging countries, a plateau has been observed for a few years in the industrialized countries with a maximum of 20% reached in Northern Europe.

The predominant symptom of AD is pruritus. It has a strong impact on the lives of patients both physically, psychologically and socially, which causes stress and sleep disorders. Because of this pruritus, sleep disturbances but also the displaying character of the disease, the quality of life of patients and their families is very often altered.

The pathophysiology of this chronic pathology and associated pruritus is complex and incompletely understood and current treatments are unfortunately only symptomatic.

Many receptors (TRPA1, TRPV1, PAR2 ...), molecules (neuromediators, neuropeptides, histamine ...) and secreted cytokines (IL-2, -4, -13 and -31, TSLP) are involved in the induction and mediation of chronic pruritus. Their role in pruritus associated with AD begins to be understood. Among them, the TRPM 8 has a particular interest. Indeed, this receptor belongs to the superfamily of the "potential transient receptor (TRP)" whose members are known to play a major role in sensory perceptions, including the perception of pruritus. TRPM8 is a thermoreceptor, activated by cold (T <28 ° C) or compounds such as menthol or derivatives, or eucalyptus and the beneficial action of menthol in the soothing of pruritus makes the TRPM8 receptor an attractive therapeutic target for treatment of pruritus in AD. Its role has never been studied in this context.

This project aims to study the role of TRPM8 in the pathophysiology of pruritus in AD in an in vitro model. Biopsies of atopic dermatitis patients (2/patient in pruritic skin lesion) will be put in culture and submit to topical application of menthoxypropanediol. The effect of this molecule on receptors involved in pruritus pathway will be assay (immunohistochemistry, QPCR).

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age with atopic dermatitis.
* AND presenting active itchy lesions,
* Patients with no systemic and / or topical treatment for AD or pruritus.
* Patients who gave their written consent

Exclusion Criteria:

* Patients with a physical or psychological disability to sign the consent.
* Patients not supported by social security.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-11-21 (Actual); Primary Completion 2019-01-29 (Actual); Study Completion 2019-01-29 (Actual)

PRIMARY OUTCOMES:
Mitigation of pruritus markers after topical application of menthoxypropanediol on AD skin biopsies : proteins expression analysis | ONE DAY
  For proteins expression analysis, Immunostaining of specific receptors and proteins will be made on skin sections of AD skin biopsy. Photos will be realized with an "Axiocam" camera and analyzed by "Axiovision" software. Staining intensity of each will be evaluated in well-defined reference areas by quantitative (immuno-)histomorphometry by using ImageJ software. Relative intensity of each receptor or protein of AD patient biopsy treated or not by menthoxypropanediol will be compared to each other and compared also to healthy skin.
Mitigation of pruritus markers after topical application of menthoxypropanediol on AD skin biopsies : transcriptomic analysis | ONE DAY
  For transcriptomic analysis, RNA from AD skin biopsies will be extracted and QPCR analysis will be performed. Variation of receptor and proteins expression with and without menthoxypropanediol treatment will be realized on AD skin and also compared to healthy skin.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Brest, Brest, France

IPD SHARING:
Plan to Share IPD: No